CLINICAL TRIAL: NCT01362166
Title: With Different Frequency Electric Signals Study the Frequency Response of the Foot-Yangming Stomach Channel: Zu-San-Li and Xian-Gu
Brief Title: Frequency Response of the Foot-Yangming Stomach Channel: Zu-San-Li and Xian-Gu
Acronym: YCFR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: China Medical University, China (Other)
Responsible Party: Institution of the Integrated Medicine, Institution of the Integrated Medicine
Other Study IDs: DMR100-IRB-034
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Healthy
Keywords: Chinese medicine; channel; acupuncture; ZuSanLi; XianGu; frequency response; resonance; male volunteer; aged within 20-35 years old

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main purpose of this study is to detect the frequency response in the electric wave transmission through the channels inside human body. With the electric signals in different frequencies, analyzed by the digital signal processing technique, the adaptability of the channel for different frequencies may be revealed. With this study there will be a feasible connection between the physiological signals and the channel theory in Chinese medicine, and the basis of the physiological signals can be drew out for the description of the internal organs, the strong or weak, the truth or falsity.

The Zu-San-Li is the open acupoint on foot-Yangming channel, the stomach channel. Qi, the main concept in TCM, will flow from the open acupoint to go into deep internal organs. Xian-Gu is another Yu acupoint on foot-Yangming channel. The inborn original Qi flows from the Yu acupoint infuse into blood vessels. So in this study the investigators will take these two acupoints for the acupuncture. Since the direction of the channel is from Zu-San-Li to Xian-Gu, the investigators pick Zu-San-Li as the input and Xian-Gu the output for the electrical signals.

For this experiment, the investigators planned enrolling 30 male sub-healthy volunteers, aged in 20-35 years old, to finish the whole experiment procedures.

After the acupuncture, the electric signals of different modes will be input from the subject's open acupoint (Zu-San-Li), and measure the frequency respond voltage from the output acupoint (Xian-Gu).

Each subject must complete the acupuncture of Zu-San-Li and Xian-Gu, and be input 5 sets of the electric signals of different modes two times on the trial. The variety conditions of the wave form and electric voltage will be recorded and measured respectively.

The investigators plan to obtain the data in six months, and complete the data analysis and sorting in two months.

ELIGIBILITY:
Inclusion Criteria:

* have never got myocardial infarction, heart failure, or any other heavy diseases
* in normal mental state, can match with the researcher
* would like to obey the experiment 24-hour related rules
* sign the written agreement

Exclusion Criteria:

* The one who has arrhythmia, or is equipped with the heart stanza machine.
* Get myocardial infarction, heart failure, and the other heavy diseases
* The mental state is unsteady.
* Female.
* Does not sign the written agreement.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-05

CONTACTS AND LOCATIONS:
Overall Officials: Fun-jou Chen, Prof., Study Director — China Medical University, China
Locations (1):
- China Medical University, Taichung, Taiwan

REFERENCES:
- [Result] Dhond RP, Yeh C, Park K, Kettner N, Napadow V. Acupuncture modulates resting state connectivity in default and sensorimotor brain networks. Pain. 2008 Jun;136(3):407-418. doi: 10.1016/j.pain.2008.01.011. Epub 2008 Mar 11. PMID 18337009
- [Result] Sakai S, Hori E, Umeno K, Kitabayashi N, Ono T, Nishijo H. Specific acupuncture sensation correlates with EEGs and autonomic changes in human subjects. Auton Neurosci. 2007 May 30;133(2):158-69. doi: 10.1016/j.autneu.2007.01.001. Epub 2007 Feb 22. PMID 17321222
- [Result] Streitberger K, Steppan J, Maier C, Hill H, Backs J, Plaschke K. Effects of verum acupuncture compared to placebo acupuncture on quantitative EEG and heart rate variability in healthy volunteers. J Altern Complement Med. 2008 Jun;14(5):505-13. doi: 10.1089/acm.2007.0552. PMID 18537467
- [Result] Napadow V, Dhond RP, Purdon P, Kettner N, Makris N, Kwong KK, Hui KK. Correlating acupuncture FMRI in the human brainstem with heart rate variability. Conf Proc IEEE Eng Med Biol Soc. 2005;2005:4496-9. doi: 10.1109/IEMBS.2005.1615466. PMID 17281236
- [Result] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210
- [Result] Guzzetti S, Piccaluga E, Casati R, Cerutti S, Lombardi F, Pagani M, Malliani A. Sympathetic predominance in essential hypertension: a study employing spectral analysis of heart rate variability. J Hypertens. 1988 Sep;6(9):711-7. doi: 10.1097/00004872-198809000-00004. PMID 3183374
- [Result] Lishner M, Akselrod S, Avi VM, Oz O, Divon M, Ravid M. Spectral analysis of heart rate fluctuations. A non-invasive, sensitive method for the early diagnosis of autonomic neuropathy in diabetes mellitus. J Auton Nerv Syst. 1987 May;19(2):119-25. doi: 10.1016/0165-1838(87)90005-1. PMID 3598051
- [Result] Axelrod S, Lishner M, Oz O, Bernheim J, Ravid M. Spectral analysis of fluctuations in heart rate: an objective evaluation of autonomic nervous control in chronic renal failure. Nephron. 1987;45(3):202-6. doi: 10.1159/000184117. PMID 3574569
- [Result] Buchman TG, Stein PK, Goldstein B. Heart rate variability in critical illness and critical care. Curr Opin Crit Care. 2002 Aug;8(4):311-5. doi: 10.1097/00075198-200208000-00007. PMID 12386491
- [Result] Cashion AK, Holmes SL, Arheart KL, Acchiardo SR, Hathaway DK. Heart rate variability and mortality in patients with end stage renal disease. Nephrol Nurs J. 2005 Mar-Apr;32(2):173-84. PMID 15889802
- [Result] Ryan C, Hollenberg M, Harvey DB, Gwynn R. Impaired parasympathetic responses in patients after myocardial infarction. Am J Cardiol. 1976 Jun;37(7):1013-8. doi: 10.1016/0002-9149(76)90417-3. PMID 1274861